CLINICAL TRIAL: NCT02312973
Title: Investigation of Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Single Oral Doses of 75 mg Molidustat in Male and Female Subjects With Renal Impairment Requiring Hemo- or Peritoneal Dialysis Compared to Age- and Weight-matched Healthy Subjects in a Single-center, Non-controlled, Non-blinded Study With Group Stratification
Brief Title: To Investigate Pharmacokinetics (Absorption, Distribution, Elimination), Safety and Tolerability of a Single Oral Dose of 75 mg Molidustat Tablet in Male and Female Subjects Requiring Hemo- or Peritoneal Dialysis Compared to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 17767; 2014-003292-31 (EudraCT Number)
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Chronic kidney disease; Pharmacokinetics; Hemodialysis; Peritoneal dialysis; Erythropoietin
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental): Single oral dose of 75 mg molidustat (fasted) in subjects on hemodialysis (at start of hemodialysis and on a hemodialysis free day,respectively)
  Interventions: Drug: Molidustat(BAY85-3934)
- Arm 2 (Experimental): Single oral dose of 75 mg molidustat (fasted) in subjects on peritoneal dialysis (after start of peritoneal dialysis intervall and, optionally, after the start of a peritoneal dialysis-free intervall,respectively)
  Interventions: Drug: Molidustat(BAY85-3934)
- Arm 3 (Experimental): Single oral dose of 75 mg molidustat (fasted) in healthy subjects
  Interventions: Drug: Molidustat(BAY85-3934)

INTERVENTIONS:
Drug: Molidustat(BAY85-3934) — Two single oral doses of 75 mg molidustat tablet in subjects on hemodialysis and peritoneal dialysis
  Arms: Arm 1; Arm 2
Drug: Molidustat(BAY85-3934) — One single oral dose of 75 mg molidustat in healthy subjects
  Arms: Arm 3

SUMMARY:
The study investigates the pharmacokinetics (absorption, distribution, elimination) of molidustat after intake of a single 75 mg tablet in subjects with renal impairment requiring hemo- or peritoneal dialysis compared to age-and gender-matched healthy subjects. In addition, the effect of molidustat on the hormone erythropoietin will be evaluated as well as the safety and tolerability of molidustat.

ELIGIBILITY:
Inclusion Criteria:

* Male and female (without childbearing potential)
* Age: ≥18 and ≤79 years of age
* Body mass index (BMI): ≥18 and ≤34 kg/m2
* Ethnicity: White
* Subjects with severe renal impairment on hemodialysis or peritoneal dialysis, and
* Healthy subjects

Exclusion Criteria:

* Women of childbearing potential, pregnant or lactating women
* Use of medication within the 2 weeks preceding the study which could interfere with the investigational product
* Positive results for hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibodies (HCV Ab), human immune deficiency virus 1 and 2 antibodies (HIV 1/2 Ab)
* Exclusion periods from other studies or simultaneous participation in other clinical studies

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01-14 (Actual); Primary Completion 2015-12-02 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics characterized by Cmax of Molidustat | Up to 96 hours post dose
  Cmax: maximum drug concentration in plasma after single dose administration
Pharmacokinetics characterized by AUC of Molidustat | Up to 96 hours post dose
  AUC: area under the plasma concentration vs time curve from zero to infinity
Pharmacokinetics characterized by Cmax,norm of Molidustat | Up to 96 hours post dose
  Cmax,norm;maximum drug concentration in plasma after single dose administration divided by dose (milligrams) per kilogram body weight
Pharmacokinetics characterized by (AUCnorm) of Molidustat | Up to 96 hours post dose
  AUCnorm; area under the plasma concentration vs time curve divided by dose per kg body weight

SECONDARY OUTCOMES:
Pharmacokinetics characterized by Cmax of erythropoietin | Up to 48 hours post dose
  Cmax: maximum drug concentration in plasma after single dose administration
Pharmacokinetics characterized by AUC (0-tlast) of erythropoietin | Up to 48 hours post dose
  AUC(0-tlast): AUC from time 0 to the last data point above lower limit of quantification
Pharmacokinetics characterized by tmax of erythropoietin | Up to 48 hours post dose
  tmax: time to reach maximum drug concentration in plasma after single (first) dose
Number of subjects with Treatment Emergent Adverse Event (TEAE) | Up to 7 days post dose

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Germany (2):
  - Velbert, North Rhine-Westphalia
  - Kiel, Schleswig-Holstein